CLINICAL TRIAL: NCT00000573
Title: Emphysema: Physiologic Effects of Nutritional Support
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized
Other Study IDs: 211; R01HL033269 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2002-04

CONDITIONS: Emphysema; Lung Diseases; Lung Diseases, Obstructive; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Emphysema; Lung Diseases; Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive | interventions — Enteral Nutrition

INTERVENTIONS:
Procedure: enteral nutrition

SUMMARY:
To determine if enteral nutrition support (ENS) restores normal body weight and improves muscle strength, exercise performance, sensation of dyspnea, and quality of life in malnourished patients with chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
BACKGROUND:

Chronic obstructive pulmonary disease is a major health problem and a leading cause for hospital admission in the United States. A severe form of chronic obstructive pulmonary disease that is accompanied by weight loss is commonly referred to as pulmonary cachexia. Studies in the 1960s demonstrated associations in chronic obstructive pulmonary disease patients between weight loss, low FEV1, and early mortality. This observation was strengthened by a retrospective analysis of the Intermittent Positive Pressure Breathing Trial data that suggested malnutrition was an independent predictor of outcome in men with chronic obstructive pulmonary disease. The underlying basis relating malnutrition to adverse outcome in chronic obstructive pulmonary disease was unknown, although there was a large body of information indicating that pulmonary cachexia was associated with respiratory muscle atrophy, myofibrillar substrate depletion, and impaired skeletal and respiratory muscle function. The primary question was whether the nutrition-related functional deficits observed in underweight patients could be reversed.

The first three years of the study supported a pilot project of oral nutrition therapy in malnourished chronic obstructive pulmonary disease patients.

DESIGN NARRATIVE:

All subjects underwent intubation during the initial testing interval and subsequently underwent dietary counseling and oral nutritional supplement during a two-month stabilization phase. Subjects who demonstrated adequate weight gain defined as achievement of more than 90 percent of ideal body weight or who were unable to tolerate intubation were eliminated from further investigation. Eligible subjects were randomized to either ENS or to dietary counseling only. Subjects randomized to ENS received enteral supplementation with Osmolite delivered by continuous infusion pump. Feedings were continuous or nocturnal for sixteen weeks in order to deliver a caloric intake of 1.7 times the resting energy value. Following the intervention phase, all subjects were maintained on dietary counseling on a monthly basis with oral nutritional supplements. Outcome variables were measured before and after the stabilization phase, at eight and sixteen weeks during the intervention phase, and at eight and sixteen weeks during the post-intervention phase. The primary outcome variable was muscle strength and its effect on exercise performance, dyspnea, and quality of life. Secondary outcome variables included morbidity and mortality. The grant was extended through November 1995 for data analysis.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
Men and women with uncomplicated stable chronic obstructive pulmonary disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1990-01; Study Completion 2005-11 (Actual)

REFERENCES:
- [Background] de Godoy I, Donahoe M, Calhoun WJ, Mancino J, Rogers RM. Elevated TNF-alpha production by peripheral blood monocytes of weight-losing COPD patients. Am J Respir Crit Care Med. 1996 Feb;153(2):633-7. doi: 10.1164/ajrccm.153.2.8564110.